CLINICAL TRIAL: NCT00721838
Title: Dietary Intake and Eating Behaviors in Adolescents Who Undergo Bariatric Surgery
Acronym: Teen LABS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Hospital Medical Center, Cincinnati (Other); Baylor College of Medicine (Other); University of Pittsburgh (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: DK072493; U01DK072493 (NIH)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Adolescent Obesity; Eating Behavior; Dietary Intake
Keywords: adolescent obesity; eating behavior; dietary intake
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Surgery group
- 2: Control - Lifestyle modification program

SUMMARY:
to study the dietary intake and eating behaviors of adolescents who undergo bariatric surgery

DETAILED DESCRIPTION:
The dietary and eating behavior outcomes for adolescents who undergo bariatric surgery are virtually unknown. The main trial of the Teen-LABS consortium is not studying dietary intake and eating behavior before and after bariatric surgery. The consortium, however, provides a unique opportunity to investigate these issues in a large and diverse sample through the context of the proposed ancillary study.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or younger
* have a BMI > 30 kg/m2
* have attained or nearly attained physical maturity and have a history of unsuccessful, organized attempts at weight management.
* must demonstrate reasonable decision making abilities
* must also fit the following criteria: (1) no prior bariatric surgical procedure, (2) no physical illness not due to obesity, and (3) no full-time special education (due to the high reading demand of study participation).
* Participants will be from all racial and ethnic groups and be both male and female.

Exclusion Criteria:

* We will not exclude participants from this trial based on health status or medication usage. Instead, we will track medical conditions and medication usage at every assessment point throughout the investigation to assess the possible influence of these variables on changes in weight, dietary intake, and eating behavior.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will assess changes in dietary intake and eating behavior in 110 extremely obese adolescents who undergo bariatric surgery as part of the main Teen-LABS study. These individuals will be recruited from one of 4 Teen-LABS sites: Baylor College of Medicine, Cincinnati Children's Hospital Medical Center, University of Alabama at Birmingham, and the University of Pittsburgh Medical Center. Changes in bariatric surgery patients will be compared to those of 110 obese adolescents treated with a lifestyle modification program designed to produce an 8% weight loss. These individuals will be recruited from a study at the Children's Hospital of Philadelphia (PI: Robert Berkowitz, M.D.) which will be ongoing at the same time and will include the same measures as those proposed in this application.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2009-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
dietary intake | BL, 3, 6, 12, and 24 mo
eating behavior | BL, 3, 6, 12, and 24 mo

SECONDARY OUTCOMES:
nausea, vomiting, and gastric dumping | BL, 3, 6, 12 and 24 mo

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The University of Pennsylvania Weight and Eating Disorder Program, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas